CLINICAL TRIAL: NCT01944592
Title: Gynaecology Teaching Associates Versus Teaching on Manikins: a Randomised Controlled Trial
Brief Title: Teaching Associates Randomised to Evaluate the Effectiveness of Gynaecological Pelvic Examination Versus Traditional Teaching Using Manikins
Acronym: TARGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Thomas Justin Clark, Consultant Obstetrician and Gynaecologist, Birmingham Women's NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: TARGET001
Record Dates: First submitted 2013-09-13; First posted 2013-09-17 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Female Pelvic Examination
Keywords: Gynaecology Teaching Associate; Pelvic examination; Students
MeSH Terms: interventions — Manikins; Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gynaecology Training Associates (GTA's) (Experimental): Final year (Year 5) medical undergraduates embarking upon their O&G clinical placement trained in pelvic examination with GTA's
  Interventions: Behavioral: Gynaecology Teaching Associates (GTA's)
- Manikin training (Active Comparator): Final year (Year 5) medical undergraduates embarking upon their O&G clinical placement trained in pelvic examination on manikins.
  Interventions: Behavioral: Manikin (conventional) training

INTERVENTIONS:
Behavioral: Gynaecology Teaching Associates (GTA's) — Two GTA's will conduct the session according to the following structure; Students will receive a short anatomy PowerPoint presentation from the GTA's followed by demonstration of a gynaecological examination on a pelvic manikin. Students will then be taken to the out-patient department where one GTA will demonstrate pelvic examination on the other. Each student will then examine one of the GTAs under supervision by the other. The three non-active students will observe each of their colleagues' examinations. The students will then undergo a role play scenario where they will examine one of the GTAs under supervision of the other and feedback will be given by both GTAs.
  Arms: Gynaecology Training Associates (GTA's)
Behavioral: Manikin (conventional) training — Clinical Lecturers in Gynaecology (equivalent to Specialist Registrar experience) will conduct the sessions as follows: Students will receive a short anatomy PowerPoint presentation (the same as used in the GTA training). The Clinical Lecturer will then demonstrate pelvic examination on the pelvic manikin. Each student will then perform the pelvic examination twice supervised by the Clinical Lecturer.
  Arms: Manikin training

SUMMARY:
Physical examination of the pelvis is an important core skill that medical students need to acquire. However, due to its intimate nature some students are graduating unable to perform competent pelvic examinations. Gynaecological Teaching Associates (GTA's) are women who have been trained to be examined and give valuable feedback to the students. In North America GTA's are quite commonly used in the medical curriculum and they have also been used in Canada, Australia and Scandinavia. In the UK pelvic examination is mainly taught using a combination of clinic patients, pelvic models and patients anaesthetised for surgery. In Birmingham we have already started using GTA's and like other Universities such as Oxford the students have given positive feedback.

GTA's are paid professionals and hence introducing this method of teaching has financial implications for Universities. Unless it is proven to be worthwhile it is unlikely that academic institutions will introduce and maintain GTA programs. One UK study did show that those who had been trained with a GTA's and pelvic models were significantly better than those who had been trained with pelvic models alone. However, in this study the GTA training was supplementary to the normal curriculum so the amount of teaching rather than the style of teaching may have acted as a confounding factor. Therefore, a large randomised trial of trainees on the Obstetrics and Gynaecology (O&G) programme comparing those given an initial teaching session on a pelvic model and those taught by GTA's is needed to assess the effectiveness of GTA's on confidence and competence of the students by the end of the training programme is needed.

DETAILED DESCRIPTION:
Introduction Physical examination of the pelvis is an important core skill that medical students need to acquire. However, the experience of undergraduates to vaginal examination is becoming increasingly limited such that medical students in Birmingham can qualify without ever performing a vaginal examination in an outpatient setting (personal communication, Raut N). It is well recognised that the intimate nature of the examination poses additional challenges to medical students and their teachers in gaining consent for supervised training. However, other factors may now be affecting student experience. These include competing pressures on contemporary undergraduate medical curricula resulting in traditional clinical placements, such as obstetrics and gynaecology (O&G), becoming shortened in many academic medical institutions. Empowerment of patients combined with changes in their expectations of interactions with medical professionals may have further restricted access to clinical cases. Changes in attitudes to teaching gynaecological examination may not be restricted to patients; medical educationalists may also have become more conservative or less experienced such that they find teaching vaginal examination an increasing challenge.

Whatever the reasons underlying the diminishing exposure of medical students to gynaecological examination are, the current status quo is unacceptable. Teaching innovations are urgently required to enhance teaching of a skill which is fundamental to both gynaecological and general medical practice. A strategy becoming increasingly popular is the use of "gynaecological teaching associates" or GTA's for short. These women are 'expert patients' who have been trained to undergo and teach gynaecological examination, giving valuable and immediate feedback to the students. In North America GTA's are quite commonly used in the medical curriculum and they have also been used in Canada, Australia and Scandinavia. In the UK pelvic examination is still mainly taught through simulation on pelvic models (manikins) combined with experience gained from supervised teaching on women attending outpatient clinics and those anaesthetised for surgery within clinical attachments. However, the length of these placements varies in length throughout UK medical schools and the quality of experience is likely to be inconsistent even within medical schools. In 2011 at the Birmingham Women's Hospital (BWH), we instituted a GTA teaching programme. Final year medical students from the University of Birmingham Medical School allocated clinical placements in O&G at the BWH undergo GTA teaching within the first week of their five week attachment. To date, in keeping with other Universities with GTA programmes experience, such as Oxford University and Kings College, London (1), our students have given universally positive feedback (Clark TJ, Personal Communication).

Anecdotal qualitative data from our students is reassuring but whether the GTA programme in its current design is effective and indeed cost-effective in key educational outcomes is unclear. The published data available are generally descriptive studies of the process and institution of GTA programmes into the undergraduate medical curriculum (2-7). Studies addressing student competence and confidence are limited to small, observational series. One non-randomised controlled study from the UK demonstrated that students who had been trained with GTA's were significantly better than those who had been trained with pelvic models alone (1). However, in this study the GTA training was supplementary to the normal curriculum so the amount of teaching rather than the style of teaching may have acted as a confounding factor. Moreover, a valid assessment tool was not used to assess clinical performance. Evaluating the educational benefit of GTAs is also important if we are to allocate scarce undergraduate educational resources efficiently. Gynaecological teaching associates are paid professionals and introducing this method of teaching has financial implications for Universities.

At present, the University of Birmingham has not fully incorporated GTA teaching into its final year O&G curriculum with 150/400 students placed at the BWH being taught in this way. Thus, with opinion as to the value of GTAs not yet solidified and in the absence of rigorous scientific assessment of the educational and economic benefits of GTAs, we propose a large randomised controlled trial. The RCT will compare the effectiveness and cost-effectiveness of teaching female pelvic examination to medical students using GTAs with traditional teaching using pelvic manikins.

Objectives

The TARGET RCT has been designed to answer the following research questions:

Principal Research Question

• Do gynaecological teaching associates improve the level of confidence of medical students in performing gynaecological pelvic examination compared to manikin based teaching?

Secondary Research question

* Do Gynaecological Teaching Associates improve the level of competence of medical students in performing gynaecological pelvic examination compared to manikin based teaching?
* Do the following factors affect the competence and confidence of medical students in performing gynaecological pelvic examination: student gender; ethnicity; perception of clinical placement; number of supervised vaginal examinations conducted during clinical placement?
* Are Gynaecological Teaching Associates cost-effective?

ELIGIBILITY:
Inclusion Criteria:

* Final year medical students
* Consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Student confidence | At the end of placement (week 5)
  At the start of the placement in O&G (during week one), the students will be asked to rate their confidence in gynaecological examination. The assessment tool comprises five questions relating to various communication and practical aspects of the procedure as well as a further global assessment of confidence. A 100mm VAS will be used to measure response. The students will be asked to rate their confidence on the same scales at the end of their placement.

SECONDARY OUTCOMES:
Student competence | At the end of placement (week 5)
  all participants will be invited to attend an assessment session under standard MB ChB examination conditions. Two senior examiners (post MRCOG specialists in Gynaecology), with an interest in Medical Education and familiarity in OSCE style assessments will assess the students independently using a validated assessment tool (Personal Communication, Clark TJ). The assessment tool comprises six domains including a global assessment with competence measured according to a 100mm visual analogue scale (VAS). The mean score over all domains will form the final student score. Examiners will be blinded to the student's group allocation.
Number of vaginal examinations performed | At the end of placement (week 5)
  The students will be asked how many vaginal examinations they have performed (excluding those on GTAs) during their five week placement under supervision on (i) women in the outpatient clinic or ward setting; (ii) women under general anaesthesia prior to operative intervention.
Student rated usefulness of training session | At the end of placement (week 5).
  All students will be asked to rate the usefulness of their initial training sessions in pelvic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Clark, MBChB MD(hons), Principal Investigator — Birmingham Women's NHS Foundation Trust
Locations (1):
- Birmingham Womens Hospital, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Pickard S, Baraitser P, Rymer J, Piper J. Can gynaecology teaching associates provide high quality effective training for medical students in the United Kingdom? Comparative study. BMJ. 2003 Dec 13;327(7428):1389-92. doi: 10.1136/bmj.327.7428.1389. PMID 14670887
- [Background] Wanggren K, Fianu Jonassen A, Andersson S, Pettersson G, Gemzell-Danielsson K. Teaching pelvic examination technique using professional patients: a controlled study evaluating students' skills. Acta Obstet Gynecol Scand. 2010 Oct;89(10):1298-303. doi: 10.3109/00016349.2010.501855. PMID 20846063
- [Background] Wanggren K, Pettersson G, Gemzell-Danielsson K. Medical students learning the pelvic examination: evaluation of a clinical patient model. Acta Obstet Gynecol Scand. 2010 Oct;89(10):1304-9. doi: 10.3109/00016349.2010.513425. PMID 20726831
- [Background] Robertson K, Hegarty K, O'Connor V, Gunn J. Women teaching women's health: issues in the establishment of a clinical teaching associate program for the well woman check. Women Health. 2003;37(4):49-65. doi: 10.1300/J013v37n04_05. PMID 12956214
- [Background] Beckmann CR, Barzansky BM, Sharf BF, Meyers K. Training gynaecological teaching associates. Med Educ. 1988 Mar;22(2):124-31. doi: 10.1111/j.1365-2923.1988.tb00422.x. PMID 3374413
- [Background] Beckmann CR, Sharf BF, Barzansky BM, Spellacy WN. Student response to gynecologic teaching associates. Am J Obstet Gynecol. 1986 Aug;155(2):301-6. doi: 10.1016/0002-9378(86)90814-8. PMID 3740146
- [Background] Plauche WC, Baugniet-Nebrija W. Students' and physicians' evaluations of gynecologic teaching associate program. J Med Educ. 1985 Nov;60(11):870-5. PMID 4057229
- [Derived] Janjua A, Roberts T, Okeahialam N, Clark TJ. Cost-effective analysis of teaching pelvic examination skills using Gynaecology Teaching Associates (GTAs) compared with manikin models (The CEAT Study). BMJ Open. 2018 Jun 22;8(6):e015823. doi: 10.1136/bmjopen-2017-015823. PMID 29934378